CLINICAL TRIAL: NCT03823755
Title: Evaluation of the Mobility of the Digital Flexor Tendons Operated by Dynamic MRI: a Pilot Study.
Brief Title: Evaluation of the Mobility of the Digital Flexor Tendons
Acronym: DynamicMRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0214
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Flexor Digitorum Longus on the Right; Flexor Digitorum Longus on the Left; Tendon Rupture; Tendon Injury - Hand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study flexor tendon excursion in the hand after surgery by dynamic MRI

DETAILED DESCRIPTION:
The study of the movement of the digital flexor tendon operated on MRI could lead to a better understanding of the biomechanics of this tendon after surgery, to objectively assess the repair of the tendon and the recovery of its mobility. The visualization of the aspect and the movement of this operated tendon would make it possible to adapt the rehabilitation for each patient and to prevent the occurrence of complications which limit functional recovery and source of handicap.

The analysis of the imaging in patients evolving would establish useful criteria the surgeon to judge the evolution of the operated tendon.

The first step consists in evaluating the feasibility of the acquisition of dynamic sequences in MRI and the possibility of observing the movement of the flexor tendon operated during the mobilization of the finger, and comparing the biomechanical data obtained with those of the nonoperated tendons and experimental models.

ELIGIBILITY:
Inclusion Criteria:

* flexor tendon injury in zone 2
* treatment by surgery
* insufficient functional outcome after surgery
* MRI requested by surgeon

Exclusion Criteria:

* pregnancy
* MRI contraindications
* previous surgery on the hand
* rheumatic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with flexor tendon injury in zone 2 and insufficient functional after surgery with MRI requested for exploration
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Flexor tendon excursion | 1 year
  Imaging of flexor tendon excursion in the hand after surgery during motion with MRI

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - Clinique Keraudren, Brest
  - HIA, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement